CLINICAL TRIAL: NCT06546683
Title: The Effect of a Short-Chain Fatty Acid Intervention on Affective Brain Circuits and Neuroepigenetics
Brief Title: Brain Responses to Short-Chain Fatty Acid Intervention
Acronym: MoodBugs HDAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lukas Van Oudenhove, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: S68154
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Stress; Healthy Volunteers
Keywords: Short-Chain Fatty Acids; Acute Stress; Microbiota-Gut-Brain-Axis; Neuroepigenetics; [11C] Martinostat; Functional magnetic resonance imaging
MeSH Terms: interventions — Fatty Acids, Volatile

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and personnel involved in data analyses are blinded to the intervention. Unblinding occurs after all data has been collected and analysed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-Chain Fatty Acids (Experimental): SCFAs will be delivered directly to the colon using pH-dependent colon delivery capsules
  Interventions: Other: Short-Chain Fatty Acids
- Placebo (Placebo Comparator): Colon-delivery capsules of microcrystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Short-Chain Fatty Acids — Colon-delivery capsules of Short-Chain Fatty Acids will be administered in a ratio of 60:20:20, thus 150 mmol of acetate, 50 mmol of propionate and 50 mmol of butyrate equivalent to 20g of fibers, once daily, one week
  Arms: Short-Chain Fatty Acids
Other: Placebo — Microcrystalline Cellulose will be used as placebo, one daily, one week
  Arms: Placebo

SUMMARY:
A randomized, triple-blind, placebo-controlled study on the effect of colon-delivered short-chain fatty acids (SCFAs) on neural responses to stress and neuroepigenetics.

DETAILED DESCRIPTION:
The goal of this interventional study is to study the underlying mechanism of the attenuating effect of colon-delivered SCFAs on the cortisol response to stress. Pre-clinical studies suggest that the histone-deacetylase (HDAC)-inhibiting properties of SCFAs are the main mechanism underlying SCFA-induced changes in stress, cognition and behavior.

Primary objective: to test the effect of colon-delivered SCFA intervention versus placebo on HDAC expression in the brain and neural responses to stress

Secondary objective: to determine the effects of colon-delivered SCFA administration versus placebo on inflammatory and autonomic responses to stress and to determine the mediating and/or moderating factors that potentially underlie SCFA-induced changes to stress responses (HDAC expression in stress-responsive regions, serum SCFA levels)

To this end, 32 participants will be asked to undergo a pre- and post-intervention visit, separated by one week intervention with either colon-delivered SCFAs or placebo (16 per group). During the study visits, participants undergo simultaneous PET-MR imaging with [11C]Martinostat. They undergo the Montreal Imaging Stress Test (MIST) and the Maastricht Acute Stress Test (MAST) at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Proficiency in English and/or Dutch
3. Access to a -18°C freezer (i.e. ordinary household freezer)
4. Male participants
5. Age 18-45 years
6. BMI 18.5-25 kg/m2

Exclusion Criteria:

1. Participant has a history of previous or current neurological, psychiatric, gastrointestinal or endocrine disorder
2. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol (as assessed by medical staff on the research team)
3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the study
4. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
5. Current or recent (3-month) medication use (especially antibiotics, cardiovascular drugs, steroids, non-steroid anti-inflammatory drugs, centrally effective drugs)
6. Current or recent (1-month) infection (e.g. common cold, influenza, COVID-19, etc.)
7. Recent (1-month) vaccination (e.g. flu shot, SARS-COV-2 vaccine, etc)
8. Smoking
9. Night-shift work
10. Adherence to special diets (e.g. vegan, vegetarian, weight-loss, lactose-free, gluten- free, etc.)
11. Use of pre- or probiotics within one month preceding the study
12. Previous experience with any of the tasks used in the study (not including questionnaires)
13. Neuroimaging contraindications
14. If the participant invokes that he does not want to be informed of eventual pathology that might be found during imaging (invokes the "right not to know")

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HDAC expression | Throughout study completion, on average 2 years
  Brain HDAC expression will be quantified using the PET radiotracer [11C]Martinostat before and after the intervention
Brain response to stress | Throughout study completion, on average 2 years
  Brain response (brain oxygenation level-dependent signals) to a fMRI-adapted stress task will be measured before and after intervention

SECONDARY OUTCOMES:
Brain metabolite concentration | Throughout study completion, on average 2 years
  Relative quantification of brain metabolites (mmol/L) using 1H-Magnetic Resonance Spectroscopy before and after intervention
Serum short-chain fatty acid levels | Throughout study completion, on average 2 years
  Quantification of serum SCFA (μM) before and after intervention
Salivary cortisol response to stress | Throughout study completion, on average 2 years
  Biological stress sensitivity is measured by quantifying cortisol levels (ng/ml) from multiple saliva samples taken before, during, and after a stress task performed during the pre-intervention and post-intervention visit
Cytokine levels | Throughout study completion, on average 2 years
  Quantification of inflammatory cytokines (pg/ml) before and after intervention
C-reactive protein levels | Throughout study completion, on average 2 years
  Quantification of hs-C-reactive protein levels (ng/ml) before and after intervention
Heart rate variability | Throughout study completion, on average 2 years
  Assessing heart rate variability (ms) with ECG before and after intervention
Blood pressure | Throughout study completion, on average 2 years
  Assessing blood pressure (systolic/diastolic mmHg) with a blood pressure monitor before and after intervention
Heartbeat | Throughout study completion, on average 2 years
  Assessing heartbeat (bpm) with a blood pressure monitor before and after intervention
Self-reported stress | Throughout study completion, on average 2 years
  Psychological stress sensitivity is measured through stress reports of the participants using the visual analogue scale (VAS). VAS scorings are taken before, during, and after a stress task performed during the pre-intervention and post-intervention visit.

OTHER OUTCOMES:
Fecal gut microbiota profile | Throughout study completion, on average 2 years
  Assessing gut microbiota profile before and after intervention
Perceived Stress Scale (PSS) | Throughout study completion, on average 2 years
  Assessing ratings on PSS. PSS scores range between 0-40 with higher scores indicating worse outcome
Gastrointestinal Symptom Rating Scale (GSRS) | Throughout study completion, on average 2 years
  Assessing ratings on the subscales of GSRS and its total score. It has 5 subscales (Reflux, Diarrhea, Constipation, Abdominal Pain, and Indigestion Syndrome). Subscale scores range from 1 to 7 and higher scores indicates a worse outcome.
Big Five Inventory 10 (BFI-10) | Throughout study completion, on average 2 years
  Measuring the Big Five personality traits, including Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness.
Generic Assessment of Side Effects | Throughout study completion, on average 2 years
  General side effects will be assessed and recorded in a structured, validated approach using the Generic Assessment of Side Effects (GASE)54. The GASE consists of 36 items asking for most frequently reported side effects for drugs based on the FDA adverse event reporting system database from all countries. Symptoms of all body parts during the last seven days will be self-reported and rated based on severity from 0 (not present) to 3 (severe).
State-Trait-Anxiety Inventory (STAI) | Throughout study completion, on average 2 years
  Assessing momentary (state) anxiety during the pre- and post-intervention visit. This inventory is part of the State-Trait Anxiety Inventory (STAI) with 20 questions specifically for state anxiety, rated on a 4-point scale. State anxiety is rated with anxiety absent and anxiety present questions. Anxiety absent questions constitute the absence of anxiety in a statement like, "I feel secure." Anxiety present questions represent the presence of anxiety in a statement like "I feel worried." The 4-point scale are as follows: 1 'not at all', 2 'somewhat', 3 'moderately so', and 4 'very much so'.
Emotion Regulation Questionnaire (ERQ) | Throughout study completion, on average 2 years
  designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression
Pittsburgh Sleep Quality Index (PSQI) | Throughout study completion, on average 2 years
  an instrument to measure the quality and patterns of sleep in adults. . It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month.
The Cognitive Assessment Questionnaire (CAQ) | Throughout study completion, on average 2 years
  to assess the frequency with which people experience cognitive failures, such as absent-mindedness, in everyday life - slips and errors of perception, memory and motor functioning. The questionnaire has 25 items which are scored from Never (0), Very rarely (1), Occasionally (2), Quite often (3) to Very often (4). A total score as well as three subscales (Forgetfulness, Distractibility, False Triggering) can be calculated.
Mainz Inventory for Microstressors (MIMIS) | Throughout study completion, on average 2 years
  retrospective assessment of microstressors over one week covering both stressor occurence and perceived stressor intensity

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, MD, PhD, Principal Investigator — KU Leuven; Annalena Fuchs, MSc, Study Director — KU Leuven; Kristin Verbeke, Pharm, PhD, Principal Investigator — KU Leuven; Boushra Dalile, PhD, Principal Investigator — KU Leuven
Locations (1):
- UZ/KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available upon publication with no time limitations.
Access Criteria: The data will be publicly available.